CLINICAL TRIAL: NCT03288194
Title: Improving Quality of Life in Outpatients With Heart Failure: A Two-arm Randomized Controlled Trial
Brief Title: Improving Quality of Life in Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-1619
Record Dates: First submitted 2017-09-15; First posted 2017-09-19 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Heart Failure; Quality of Life
MeSH Terms: conditions — Heart Failure | interventions — Time Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Problem-Solving Treatment (Experimental): Problem-Solving Treatment is a structured, yet flexible, form of cognitive-behavioral psychotherapy intended to increase problem-solving skills.
  Interventions: Behavioral: Problem-Solving Treatment
- Time Management (Active Comparator): Time Management is a structured, yet flexible, intervention intended to increase creativity.
  Interventions: Behavioral: Time Management

INTERVENTIONS:
Behavioral: Problem-Solving Treatment
  Arms: Problem-Solving Treatment
Behavioral: Time Management
  Arms: Time Management

SUMMARY:
This research study has been designed to test the efficacy of telephone-delivered Problem-Solving Treatment (PST) for improving the quality of life (QoL) in outpatients with stable heart failure (HF).

DETAILED DESCRIPTION:
Heart failure (HF) is the end stage of all cardiovascular diseases, and it imposes a huge burden in the United States in terms of morbidity, mortality, and economic cost. Although disease management programs have been developed to curb these costs and address the complexities of HF management, evaluations of these programs have yielded equivocal results.

With this study the Investigators plan to: (1) to determine the feasibility of telephone delivered PST for outpatients with HF and reduced QoL by obtaining estimates of yield, retention, patient acceptance, and patient satisfaction; (2) to determine whether telephone-delivered PST is associated with greater improvements in QoL than telephone-delivered Time Management over 8 weeks; and (3) to determine whether telephone-delivered PST is associated with greater reductions in depressive symptoms and/or greater improvements in self-efficacy or objectively assessed daily physical activity than telephone-delivered Time Management over 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient
* Age > 21
* Exhibits symptoms of hear failure (NYHA Class II or III)
* Left ventricular ejection fraction (LVEF) >= 40%
* Kansas City Cardiomyopathy Questionnaire (KCCQ) summary score < 60

Exclusion Criteria:

* Cannot speak English
* Lack telephone access
* Unwilling to be randomized, or
* Unavailable for the study period
* Awaiting a heart transplant (United Network for Organ Sharing Status 1A or 1B), or
* Planned (within 6 months) cardiac surgery
* Cognitive impairment indicative of dementia
* Recent (3 months)

  * acute myocardial infarction,
  * cardiac decompensation, or
  * HF-related hospitalization.
* Use intravenous inotropic medication
* Use an assistive circulatory device
* Significantly reduced life expectancy due to co-morbidity (e.g., malignancy)
* Currently receiving mental health counseling;
* A history of:

  * bipolar disorder,
  * psychosis, or
  * substance abuse/dependency
* Severe depressive symptoms or suicidality

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-04-24 (Actual); Study Completion 2017-04-24 (Actual)

PRIMARY OUTCOMES:
Change in Kansas City Cardiomyopathy Questionnaire | 1 month, 2 months, 3 months, 4 months, 5 months
  The Kansas City Cardiomyopathy Questionnaire is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life.

SECONDARY OUTCOMES:
Change in Beck Depression Inventory | 1 month, 2 months, 3 months, 4 months, 5 months
  The Beck Depression Inventory is a 21-question multiple-choice self-report inventory, one of the most widely used psychometric tests for measuring the severity of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan A Shaffer, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided